CLINICAL TRIAL: NCT00331201
Title: SAFEstart Treatment for NICU Patients With Feeding Intolerance; a Phase II Randomized, Controlled Trial
Brief Title: SAFEstart Feeding Intolerance Study Phase II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 402
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-11

CONDITIONS: Feeding Intolerance; Abdominal Distention; Gastric Residual; Emesis and Diarrhea; Blood in Stool
Keywords: NEC
MeSH Terms: conditions — Vomiting; Diarrhea; Gastrointestinal Hemorrhage

INTERVENTIONS:
Drug: SAFEstart

SUMMARY:
Feeding intolerance is a common problem in the NICU. Feeding intolerance complicates the hospitalization, lengthens the hospital stay, and adds substantially to the cost of care. We developed a method aimed at treating intestinal villous atrophy. We accomplished preclinical testing of the product, and four Phase I clinical trials, including two at McKay-Dee Hospital in 2004. Our preparation is a sterile, isotonic, solution that simulates human amniotic fluid in electrolyte composition, albumin concentration, and two enterocyte growth factors that are present in human amniotic fluid; erythropoietin and granulocyte colony-stimulating factor. We termed the product SAFEstart, using the acronym Simulated Amniotic Fluid for Enteral administration. This trial on the efficacy and safety of SAFEstart administration as a treatment for neonates who have feeding intolerance.

Hypothesis is that infants with feeding intolerance, randomized to the SAFEstart will have a greater enteral calories per kilogram per day for the seven days following conclusion of the SAFEstart administration.

DETAILED DESCRIPTION:
Feeding intolerance is relatively common in the NICU. It can manifest as emesis, diarrhea, increased abdominal girth (bloating), or in the most severe cases as necrotizing enterocolitis. Feeding intolerance complicates the hospitalization, lengthens the hospital stay, and adds substantially to the cost of care. Feeding intolerance likely has many causes. One cause that may be particularly common in the NICU is atrophy of the intestinal mucosa, which occurs during enteral fasting (when a patient is NPO). Significant intestinal villous atrophy occurs after being NPO for even 1-2 days; even if parenteral nutrition is adequate.

We developed a method aimed at preventing intestinal villous atrophy of neonates who are NPO. We accomplished preclinical testing of the product, and we completed two Phase I clinical trials involving 60 neonates. Our preparation is a sterile, isotonic, solution that simulates human amniotic fluid in electrolyte composition, albumin concentration, and two enterocyte growth factors that are present in human amniotic fluid; erythropoietin and granulocyte colony-stimulating factor. We termed the product SAFEstart, using the acronym Simulated Amniotic Fluid for Enteral administration.

SAFEstart has been tested in neonates who have never been fed, as a means of preventing villous mucosal atrophy. However, it has not yet been tested in neonates who develop feeding intolerance after several days or weeks of life. When feeding intolerance develops in such patients, the current treatments include changing formulas, continuous feeding, but does not include using SAFEstart.

It is possible that SAFEstart administration, 2.5 mL/kg enterally every three hours as we have previously done with preterm neonates beginning on the first day of life, would provide benefit to these older neonates with acquired feeding intolerance. If such infants have mucosal atrophy as part of their feeding problem, the growth factors in SAFEstart might indeed result in improved feeding tolerance.

We propose a Phase II exploratory trial among 20 neonates in the McKay-Dee NICU who develop the problem of feeding intolerance. Specifically, we propose that when feeding intolerance is diagnosed, 20 mL/kg/day of SAFEstart will be administered (every three hour gavage or nipple feedings) and that this will be continued for a period of up to one week, in an attempt to resolve the feeding intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Have feeding intolerance (defined in the following section).
* Be expected (by declaration of the Attending Neonatologist) to survive at least 28 days.
* Have documented informed consent for participation in the study.

Exclusion Criteria:

* Have a congenital surgical condition involving the intestine, such as tracheoesophageal fistulae, diaphragmatic hernia, Hirschprung's disease, bowel atresia, gastroschisis, or omphalocele.
* Be so ill as to require mechanical ventilation with >50% FIO2 at the time of study entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2005-07; Study Completion 2006-04

PRIMARY OUTCOMES:
The primary outcome measure will be the number of calories/kg taken enterally during the seven days after the four days of SAFEstart (or sham) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cindy K Barney, NNP, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- McKay-Dee Hospital Center, Ogden, Utah, United States